CLINICAL TRIAL: NCT00324506
Title: A Randomized, Open-label, Parallel-Group Multicenter Study to Determine the Safety/Efficacy of Mycophenolate Mofetil in Mono & Combination Therapy With Interferon Beta 1a in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Safety and Efficacy of Cellcept and Avonex as Combination Treatment in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Aspreva Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Elliot Frohman, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT 355349; IRB #012006-028
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cellcept and Avonex (Active Comparator)
  Interventions: Drug: Mycophenolate Mofetil (CellCept)

INTERVENTIONS:
Drug: Mycophenolate Mofetil (CellCept)

SUMMARY:
The primary objective of this safety/mechanistic study is to determine the safety and tolerability of oral Cellcept when compared with weekly intramuscular Avonex in relapsing multiple sclerosis. Safety will be assessed by virtue of changes in size and number of lesions on MRI scans.

DETAILED DESCRIPTION:
Sixty patients (20 patients at each recruiting center) with RR MS who satisfy both inclusion and exclusion criteria will be treated with CellCept® or Avonex® for the first 6 months of the study. Those patients will have a fifty-fifty chance of receiving either Avonex or Cellcept. Baseline data will be collected before treatment begins including MRIs, chest x-ray, EKG, and standard labwork, along with a blood test for HIV and Hepatitis B. Once enrolled, study visits include periodic MRI scans, a neurological exam by the examining neurologist every three months, frequent bloodwork, questionnaires, and eye-testing at month zero, six, and twelve months. Eye testing takes about one hour and requires dilation of pupils. All assessments are standard of care for ophthalmology with the exception of optical coherence tomography (OCT)-- a non-invasive procedural device that records graphical and numerical measurements of the optic nerve and macula.

All patients will begin active combination therapy on both CellCept® and Avonex® during the second 6 months of the study. During this second phase, MRI and clinical examinations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with clinically definite MS according to McDonald criteria #1-#4
* Age 18-55
* Have a RR disease course
* Have EDSS scores less than or equal to 5.0
* Have a disease duration of one day to 20 years
* Have at least one medically documented clinical relapse within the 12 months prior to randomization (for eligibility, a pre-study relapse will be defined as neurologic symptoms and signs documented by review of the history with the subject or in the medical record, of sufficient severity and duration to be determined by the investigator as consistent with an acute MS relapse; the relapse does not need to have been treated to qualify) and/or have progression of ≥1.0 points in EDSS in the previous year
* Have ≥1 Gd-enhancing brain lesion on a monthly run-in baseline MRI and ≥2 T2 brain lesions consistent with MS on the screening scan
* Signed informed consent
* None of the exclusion criteria

Exclusion Criteria:

* Previous treatment 3 months prior to study entry with standard disease-modifying therapy (interferon-beta and glatiramer acetate, IVIG and plasmaphoresis).
* Previous treatment 12 months prior to study entry with immunosuppressant agents, e.g., mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine or total body irradiation or any other concomitant immunomodulatory therapies (e.g., azathioprine, methotrexate,, CellCept®, natalizumab, and other immunomodulators/monoclonal agents).
* Patients who received steroid treatment 30 days prior to the MRI scan date
* Women who are pregnant, lactating or of childbearing age who do not consent to approved contraceptive use during the study.
* Abnormal blood tests, performed during the screening visit (see adverse events section)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2006-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this safety/mechanistic study is to determine the safety and tolerability of oral Cellcept when compared with weekly intramuscular Avonex in relapsing multiple sclerosis. Safety will be assessed by virtue of changes in MRI | 1 year

SECONDARY OUTCOMES:
Secondary Objectives: | one year
Changes in exacerbation frequency, incidence of exacerbations in the treated groups, changes in level of sustained disability | one year
, changes in quality of life measures, assessment of fatigue | one year

CONTACTS AND LOCATIONS:
Overall Officials: Elliot M Frohman, MD/PhD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (3):
- United States (3):
  - Michigan Institute for Neurological Disorders (M.I.N.D.), Farmington Hills, Michigan
  - Buffalo Neuroimaging Analysis Center (BNAC), Buffalo, New York
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas